CLINICAL TRIAL: NCT06010459
Title: Determination of 6 Minute Pegboard and Ring Test Exercise Test Reference Values in for the Turkish Healthy Adults
Brief Title: Reference Values for the Six-minute Pegboard and Ring Test in Healthy Adults in Turkey
Status: Completed | Type: Observational
Sponsor: Ulaş Ar (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Sponsor-Investigator, Ulaş Ar, Investigator, Ankara City Hospital Bilkent
Organization: Ankara City Hospital Bilkent (Other)
Other Study IDs: PBRT
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Exercise Tolerance
Keywords: Upper extremity exercise test; six-minute peg board and ring test; exercise tolerance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Supported or unsupported arm activities are widely used in all activities of daily living. 6 PBRT is a valid, reliable, useful, practical and easy-to-apply test that evaluates unassisted arm endurance in patients with COPD, asthmatics, and healthy individuals. Studies have recently been conducted showing reference values for 6 PBRT in various populations. 6 Normative values and reference range for PBRT are not available for various ethnicities, including the Turkish population. Therefore, this study aimed to find reference values for 6 PBRT in the Turkish young and middle-aged individuals.

DETAILED DESCRIPTION:
Supported or unassisted arm activities are widely used for all activities of daily living. They contribute greatly to performing both simple and complex daily tasks such as brushing, shaving, combing their hair, washing dishes or putting food on shelves; meanwhile, trapezius, pectoralis minor, scalene and intercostal muscles assist arm positioning.

Many studies; It has confirmed that patients with COPD have reduced arm exercise capacity and often experience notable dyspnoea (shortness of breath) and fatigue during arm tasks important to daily living. Two mechanisms have been suggested underlying this: neuromechanical dysfunction of the respiratory muscles (diaphragm and accessory respiratory muscles) (thoracoabdominal asynchrony) and changes in lung volume during activities involving the upper extremities. During arm exercise, accessory respiratory muscles are used for arm function and cannot contribute to respiration. This increases the respiratory load of the mechanically disadvantaged diaphragm and results in thoracoabdominal synchrony and severe dyspnea. Since the muscles that move the arm and stabilize the trunk are attached to the rib cage, they increase the resistance of the chest wall and limit the ability to increase tidal volume during arm activities. These disturbances in ventilatory mechanics result in termination of arm exercise in patients with COPD at lower workloads compared to healthy subjects.

The '6 Minute Pegboard and Ring Test-6PRT' is a valid and reliable, useful, practical and easy-to-apply test that evaluates unassisted arm endurance in COPD patients, asthmatic patients and healthy individuals. For the test, patients are asked to carry as many rings as possible within 6 minutes and the number of rings carried during 6 minutes is recorded as a score.

In a study conducted in patients with mild to very severe COPD, a positive correlation was shown between the 6PRT score and the activity counts evaluated by accelerometer. In addition, it was determined that the 6PRT score showed a clear relationship with the upper extremity ADL, and it was concluded that the 6PRT test could be used as an appropriate test for estimating and demonstrating the improvement of ADL in pulmonary rehabilitation programs.

Studies have recently been published showing reference values for 6PBRT in Brazilian and Indian populations. In one of the results, a correlation was found between the score value and age, showing that younger individuals were able to move more rings than the older group. In addition, a weak correlation was found between the test score and the level of physical activity. Normative values and reference range for 6PBRT are not available for various ethnicities, including the Turkish adults. Therefore, in this study; It is aimed to find reference values for the 6PBRT test in the Turkish adults.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 20-65 years,
* Volunteering to participate in the research
* To be cooperative
* Being between 18.5-40 kg/m2 according to body mass index value

Exclusion Criteria:

* Having a neurological disease or other clinical diagnosis that may affect cognitive status,
* Having a musculoskeletal, neurological, cardiopulmonary, neuromuscular or metabolic disease that may affect exercise performance, or having an advanced orthopedic disease (such as kyphoscoliosis),
* Recent shoulder or thoracic surgery.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy people aged 20-65 years
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Unsupported Arm Exercise Capacity and Arm Function/Endurance | 50 minute
  It will be evaluated with the '6 minute Pegboard and Ring Test-6PRT'. During the test, the patient is asked to sit in front of a pegboard and move as many rings as possible from the two lower holes to the two upper holes, using both hands simultaneously, for 6 minutes. Before the test, participants get used to the test by wearing a few rings. Standardized encouragement is given every minute during the test. The number of rings carried during 6 minutes constitutes the final score. Before and after the test, heart rate and oxygen saturation with pulse oximetry, dyspnea, general fatigue and arm fatigue perception with modified Borg scale are questioned. For the validity of the test, the test will be repeated in the same patient with one week intervals under the same conditions.

SECONDARY OUTCOMES:
Arm length of both sides and the arm and forearm circumferences of the dominant arm | 1 day
  The measurement was done with non-stretch tape
Physical Activity Level | 1 day
  It was evaluated with the Human Activity Profile.The level of physical activity of individuals is classifi ed by calculating the adjusted activity score (AAS), resulting in their being classifi ed as inactive or debilitated (AAS < 53 points), moderately active (AAS between 53 and 74 points), or active (AAS > 74 points)

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Calik Kutukcu, Assoc.Prof., Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe Üniversitesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No